CLINICAL TRIAL: NCT01365260
Title: A Double-Blind, Randomized, Feasibility Controlled Study to Assess the Safety and Efficacy of MM-II, an Injectable Intraarticular Medical Device, Intended to the Treatment of Symptomatic Knee Osteoarthritis
Brief Title: Safety and Efficacy of an Injectable Medical Device to Treat Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moebius Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM-002; 0196-11-HMO (Other: Hadassah Medical Center); HTA 5960 (Other: Israel Ministry of Health)
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MM-II (Experimental)
  Interventions: Device: MM-II
- DurolaneTM (Active Comparator): hyaluronic acid
  Interventions: Device: DurolaneTM

INTERVENTIONS:
Device: MM-II — Single intraarticular (knee) injection of MM-II
  Arms: MM-II
Device: DurolaneTM — Single intraarticular (knee) injection of DurolaneTM
  Other Names: hyaluronic acid
  Arms: DurolaneTM

SUMMARY:
The purpose of this study is to determine whether MM-II is effective in the treatment of osteoarthritis, in direct comparison with an approved hyaluronic acid preparation.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the commonest form of joint disease, characterized by articular cartilage degradation with an accompanying periarticular bone response and a synovial membrane inflammation. Clinical manifestations of OA in the knee include pain in and around the joint, stiffness of the joint after rest, crepitus on motion and limited joint. MM-II medical device was designed to reduce wear and lower friction in knees of osteoarthritis patients by creating a lubricating layer onto cartilage surfaces upon injection. The purpose of this study is to determine whether a medical device MM-II is effective in the treatment of osteoarthritis, in direct comparison with an approved hyaluronic acid preparation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic unilateral knee tibiofemoral OA
* Radiographic evidence of knee OA of Kellgren-Lawrence Grade II or III in one or both knees on a recent 3 months time X-Ray
* Knee pain within the last 24 hours before assessment more than 40mm on VAS
* Pain on most days in the last month

Exclusion Criteria:

* Knee pain equal or more than 80mm on a 100mm VAS.
* Pain in the contra lateral knee; more than 30mm on a 100 VAS.
* Concomitant inflammatory joint disease (e.g. gout, rheumatoid arthritis, history of Reiter's syndrome, psoriatic arthritis and ankylosing spondylitis.
* Any condition that may interfere with the measure of pain in the targeted knee
* Concomitant meaningful synovial fluid effusion
* Post trauma OA
* Gross ligamentous instability of the knee

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with an acute inflammatory reaction in the injected knee | up to 7 days
  An acute inflammatory reaction in more than 5% of the participants will be considered as manifestation of treatment related intolerance
Change from baseline in blood count | 3 days and 7 days
Number of participants with adverse events | Up to 90 days after the treatment

SECONDARY OUTCOMES:
Maximum global pain in the target knee | Days -21, 0, 1, 3, 7, 14, 30, 90th
  Measured by Visual Analogue Scale for pain (VAS)
The Western Ontario and McMaster University OA index (WOMAC) | Days 0, 7, 14, 30, 90
The patient global assessment of treatment by Likert-scale questionnaire | Days 0, 7, 14, 30, 90
The patients acceptance of symptoms state (PASS) | Days 7, 14, 30, 90
Omeract-ORASI responders index | Days 7, 14, 30
The number of tablets of rescue medications used between visits | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Leonid (Arieh) Kandel, MD, Principal Investigator — Hadassah Mount Scopus Hospital
Locations (1):
- Hadassah Mount Scopus Hospital, Jerusalem, Israel